CLINICAL TRIAL: NCT01248975
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Three-Treatment, Three 6-Week Period Cross-Over, Multi-Center Study to Evaluate the Effect of Adding GSK2190915 300mg as Compared to Adding Montelukast 10mg or Placebo Tablets QD to Fluticasone Propionate/Salmeterol 250/50mcg Diskus BID
Brief Title: Safety and Efficacy Study Adding GSK2190915 to Mid-dose Inhaled Corticosteroid/Long Acting Beta Agonist Combination Treatment for Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 114387
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: asthma; GSK2190915
MeSH Terms: conditions — Asthma | interventions — BID protein, human; 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- FP/SAL 250/50mcg BID plus GSK2190915 300mg QD (AM) (Experimental): FP/SAL 250/50mcg BID plus GSK2190915 300mg QD (AM)
  Interventions: Drug: FP/SAL 250/50mcg BID; Drug: GSK2190915 200mg QD (AM); Drug: GSK2190915 100mg QD (AM); Drug: Placebo capsule (PM)
- FP/SAL 250/50mcg BID plus montelukast 10mg QD (PM) (Active Comparator): FP/SAL 250/50mcg BID plus montelukast 10mg QD (PM)
  Interventions: Drug: FP/SAL 250/50mcg BID; Drug: Montelukast 10mg QD (PM); Drug: Placebo tablets (2) (AM)
- FP/SAL 250/50mcg BID plus placebo BID (Placebo Comparator): P/SAL 250/50mcg BID plus placebo BID
  Interventions: Drug: FP/SAL 250/50mcg BID; Drug: Placebo tablets (2) (AM); Drug: Placebo capsule (PM)

INTERVENTIONS:
Drug: FP/SAL 250/50mcg BID — FP/SAL 250/50mcg BID
Drug: GSK2190915 200mg QD (AM) — GSK2190915 200mg QD (AM)
  Arms: FP/SAL 250/50mcg BID plus GSK2190915 300mg QD (AM)
Drug: GSK2190915 100mg QD (AM) — GSK2190915 100mg QD (AM)
  Arms: FP/SAL 250/50mcg BID plus GSK2190915 300mg QD (AM)
Drug: Montelukast 10mg QD (PM) — Montelukast 10mg QD (PM)
  Arms: FP/SAL 250/50mcg BID plus montelukast 10mg QD (PM)
Drug: Placebo tablets (2) (AM) — Placebo tablets (2) (AM)
  Arms: FP/SAL 250/50mcg BID plus montelukast 10mg QD (PM); FP/SAL 250/50mcg BID plus placebo BID
Drug: Placebo capsule (PM) — Placebo capsule (PM)
  Arms: FP/SAL 250/50mcg BID plus GSK2190915 300mg QD (AM); FP/SAL 250/50mcg BID plus placebo BID

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of adding GSK2190915 300mg or placebo tablets administered once daily to fluticasone propionate/salmeterol 250/50mcg inhalation powder administered twice daily in uncontrolled asthmatic subjects > or = 18 years of age over the course of 6 weeks treatment.

The secondary objectives are to undertake an exploratory analysis of the efficacy and safety of adding montelukast 10mg administered once daily to fluticasone propionate/salmeterol 250/50mcg inhalation powder administered twice daily and to investigate the pharmacokinetics and pharmacodynamics of GSK2190915 in uncontrolled asthmatic subjects > or = 18 years of age over the course of 6 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years of age or older
* Non-, former or current smokers with a documented smoking history of ≤ 10 pack years
* Asthma diagnosis as defined by the National Institutes of Health
* Best FEV1 of 50% to <80% of the predicted normal value
* For current and former smokers, a post-albuterol FEV1/FVC ratio of >0.70 at Visit 1/1a (between 5:00AM and 12:00 noon)
* ≥ 12% and ≥200mL reversibility of FEV1
* Must have been using FP/SAL 250/50mcg inhalation powder BID for at least 2 weeks just prior to Visit 1.
* Must be able to replace their current short-acting beta2-agonists with albuterol inhalation aerosol
* Must be able and willing to give written informed consent to take part in the study.
* Must be able and willing to comply with all aspects of the study including completion of daily e-Diary.

Exclusion criteria:

* History of life-threatening asthma
* Recent asthma exacerbation
* Concurrent respiratory disease
* Recent respiratory infection
* Liver disease
* Other concurrent diseases/abnormalities
* Oral candidiasis
* Drug allergy
* Milk protein allergy
* Immunosuppressive Medications
* Administration of systemic, oral or depot corticosteroids within 12 weeks of Visit 1
* OATP1B1 substrates within 4 weeks of Visit 1
* Cytochrome P450 3A4 (CYP 3A4) Inhibitors
* Cytochrome P450 3A4 (CYP 3A4) Inducers
* Investigational Medications
* Compliance: any infirmity, disability, or geographical location which seems likely (in the opinion of the Investigator) to impair compliance with any aspect of this study protocol
* Affiliation with Investigator's Site

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Trough (AM pre-dose and pre-rescue bronchodilator) FEV1 | at the end of the 6 week treatment period.

SECONDARY OUTCOMES:
• Daily trough (AM pre-dose and pre-rescue bronchodilator) AM PEF | averaged over the last 3 weeks of the 6 week treatment period.
• Daily PM PEF | averaged over the last 3 weeks of the 6 week treatment period.
• Daily (average of AM and PM) | averaged over the last 3 weeks of the 6 week treatment period
• Daily asthma symptom score | averaged over the last 3 weeks of the 6 week treatment period.
• Daily rescue salbutamol use | averaged over the last 3 weeks of the 6 week treatment period.
• Percentage of symptom-free days | during the last 3 weeks of the 6 week treatment period.
• Percentage of symptom-free nights | during the last 3 weeks of the 6 week treatment period.
• Percentage of rescue-free days | during the last 3 weeks of the 6 week treatment period.
• Percentage of rescue-free nights | during the last 3 weeks of the 6 week treatment period.
• Percentage of nights without awakenings due to asthma | during the last 3 weeks of the 6 week treatment period.
• Proportion of subjects withdrawn due to lack of efficacy | during the last 3 weeks of the 6 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Bulgaria (3):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Varna
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Tarnów
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Snowise NG, Clements D, Ho SY, Follows RM. Addition of a 5-lipoxygenase-activating protein inhibitor to an inhaled corticosteroid (ICS) or an ICS/long-acting beta-2-agonist combination in subjects with asthma. Curr Med Res Opin. 2013 Dec;29(12):1663-74. doi: 10.1185/03007995.2013.842163. Epub 2013 Sep 19. PMID 24010736
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register